CLINICAL TRIAL: NCT06951984
Title: Hydroxyephedrine PET/CT in Sympathetic Nervous System Diseases
Brief Title: Hydroxyephedrine PET/CT in Sympathetic Nervous System Disease
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University (Other)
Collaborators: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Shaobo Yao, PhD, Prof., Tianjin Medical University
Other Study IDs: TJMUGH-10
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Sympathetic Nervous System Diseases; Sympathetic Nervous Structure Injury; Sympathetic Nerve Injury
Keywords: PET/CT; MRI; Hydroxyephedrine
MeSH Terms: conditions — Autonomic Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group Assignment: Each subject receive a single intravenous injection of 11C/18F-HED and undergo PET/CT or MRI imaging within the specificed time.
  Interventions: Diagnostic Test: 11C/18F-HED

INTERVENTIONS:
Diagnostic Test: 11C/18F-HED — Each subject receive a single intravenous injection of 11C/18F-HED and undergo PET/CT or MRI imaging within the specificed time.

SUMMARY:
To evaluate the potential usefulness of 11C/18F-HED positron emission tomography/ computed tomography (PET/CT) for the diagnosis of primary and metastatic lesions in various Tau-related disease patients.

DETAILED DESCRIPTION:
Subjects with various sympathetic nerves-related disease patients underwent 11C/18F-HED PET/CT either for an initial assessment or for recurrence detection. Lesions uptake was quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 11C/18F-HED PET/CT were calculated.

ELIGIBILITY:
Inclusion Criteria:

* (i) adult patients (aged 18 years or order); (ii) patients with suspected or new diagnosed or previously treated malignant tumors (supporting evidence may include MRI, CT, tumor markers and pathology report); (iii) patients who had scheduled HED PET/CT scan; (iv) patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

* (i) patients with non-malignant lesions; (ii) patients with pregnancy; (iii) the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: (i) adult patients (aged 18 years or order); (ii) patients with suspected or new diagnosed or previously treated malignant tumors (supporting evidence may include MRI, CT, tumor markers and pathology report); (iii) patients who had scheduled HED PET/CT scan; (iv) patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-03-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) | 30 days
  Standardized uptake value (SUV) of 11C/18F-HED for each target lesion of subject or suspected primary tumor or/and metastasis.

SECONDARY OUTCOMES:
Diagnostic efficacy | 30 days
  The sensitivity, specificity and accuracy of HED PET/CT were calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No